CLINICAL TRIAL: NCT00004899
Title: Autologous Bone Marrow Transplantation for Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome - A Phase II Pilot Study
Brief Title: Chemotherapy Plus Bone Marrow Transplantation and Filgrastim in Treating Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 91H1T; NU-91H1T; NCI-G00-1688
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute promyelocytic leukemia (M3); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute erythroleukemia (M6); secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b); previously treated myelodysplastic syndromes; myelodysplastic/myeloproliferative disease, unclassifiable; atypical chronic myeloid leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Congenital Abnormalities | interventions — Filgrastim; Busulfan; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: etoposide
Procedure: autologous bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing and die. Bone marrow transplantation may be able to replace cells that were destroyed by chemotherapy. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus bone marrow transplantation and filgrastim in treating patients who have acute myelogenous leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall survival and disease free survival of patients with acute myelogenous leukemia or myelodysplastic syndrome treated with busulfan and etoposide followed by autologous bone marrow transplantation and filgrastim (G-CSF).
* Assess the toxicities of this regimen in this patient population.
* Assess the hematologic effects and toxicities of G-CSF given in this setting to these patients.
* Determine whether G-CSF stimulates leukemic relapse in these patients.
* Determine whether G-CSF has an affect on platelet recovery in this setting in these patients.

OUTLINE: Patients are stratified according to first, second, or third remission. Patients undergo bone marrow collection.

Patients receive oral busulfan every 6 hours for 16 doses on days -5, -4, -3, and -2. Patients receive etoposide IV over 4 hours on days -4, -3, and -2. Bone marrow is reinfused 36-48 hours after the last dose of etoposide. Patients receive filgrastim (G-CSF) IV daily beginning 2-4 hours after bone marrow reinfusion until hematopoietic recovery.

Patients are followed monthly for 1 year, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically proven (from bone marrow aspirate smears or touch preps of marrow biopsy) of myelodysplastic syndrome or acute myelogenous leukemia (AML) of 1 of the following subtypes:

  * Acute myeloblastic leukemia (FAB M1 or M2)
  * Acute promyelocytic leukemia (FAB M3)
  * Acute myelomonocytic leukemia (FAB M4)
  * Acute monocytic leukemia (FAB M5)
  * Acute erythroleukemia (FAB M6)
* In complete remission at time of marrow or stem cell harvesting
* No relapsed AML unless bone marrow or peripheral blood stem cells previously harvested in remission are available for transplantation
* May have had secondary AML that is either therapy related or that has evolved from an antecedent myelodysplastic syndrome
* History of CNS disease during induction allowed provided inactive and cytologic examination of spinal fluid from preharvest lumbar puncture shows no evidence of leukemia
* No occult or symptomatic leukemic meningitis during induction therapy or prior to bone marrow harvesting

PATIENT CHARACTERISTICS:

Age:

* Physiologic 65 and under

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* Cardiac ejection fraction normal

Pulmonary:

* FEV1 at least 60% predicted
* DLCO at least 60% predicted

Other:

* HIV negative
* No evidence of persistent infections
* No concurrent organ damage or medical problems that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent antibiotics

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Tallman, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States